CLINICAL TRIAL: NCT04251728
Title: Acute and Chronic Effects of Automated Mechanical Peripheral Stimulation on Cardiovascular Variables in Patients With Parkinson's Disease
Brief Title: Effects of AMPS on Cardiovascular Variables in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Principal Investigator, Antonio Roberto Zamunér, Adjunct Professor - Principal Investigator, Universidad Católica del Maule
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 183/2018
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, two-arm, parallel-group study
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be assigned to Exercise plus AMPS group or Exercise plus Placebo. The placebo consist in replicating the same experimental setting and procedure, but the intensity of the stimulus is not sufficient to elicit an effect.
  The outcomes assessor will be in charge only of the evaluations with no information about the group participants belong to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise plus AMPS group (AMPS-G) (Experimental): Physical exercise and automated mechanical peripheral stimulation (AMPS) with intensity at the pain threshold, performed two times a week for 12 weeks.
  Interventions: Device: Automated mechanical peripheral stimulation; Other: Physical Exercise
- Exercise plus SHAM group (Exercise-G) (Sham Comparator): Physical exercise and simulated automated mechanical peripheral stimulation (AMPS) with intensity at the sensory threshold performed two times a week for 12 weeks.
  Interventions: Other: Physical Exercise; Device: SHAM

INTERVENTIONS:
Device: Automated mechanical peripheral stimulation — Automated mechanical pressure reaching the pain threshold in four specific points at the foots soles
  Other Names: Mechanical somatosensory stimulation; Gondola
  Arms: Exercise plus AMPS group (AMPS-G)
Other: Physical Exercise — The exercise program will be conducted for 12 weeks lasting 1 hour each session. Sessions will be held in groups and each session will comprise 4 steps: 1) Warm-up (5 min): patients will perform stretching of the main muscle groups of upper limbs, lower limbs and trunk; 2) Aerobic exercise (30 min): patients will perform continuous aerobic exercise consisting of walk on flat ground and ramps; 3) Resistance exercise training (20 min): volunteers will perform resistance exercises (2 sets x 15 repetitions) for upper and lower limbs, and trunk working the following muscle groups: shoulder flexors, extensors and abductors; elbow flexors and extensors; trunk extensors and flexors; knee flexors and extensors; and dorsiflexors and plantar flexors; 4) Cool-down (5 min): Stretching of the main muscle groups worked during the sessions and relaxation.
  Other Names: Exercise; Aerobic exercise
Device: SHAM — Automated mechanical pressure reaching the sensory threshold in four specific points at the foots soles
  Arms: Exercise plus SHAM group (Exercise-G)

SUMMARY:
This study evaluates the addition of automated mechanical peripheral stimulation (AMPS) to physical exercise in the treatment of cardiovascular and motor disabilities in Parkinson's patients. Half of participants will receive AMPS and exercise, while the other half will receive a simulated session (SHAM) and exercise.

DETAILED DESCRIPTION:
Cardiovascular abnormalities are frequent in Parkinson's disease (PD) even in the early stages. As consequence, patients may experience orthostatic hypotension and/or arterial hypertension in the supine posture, especially at night. Thus, the management of dysautonomia in patients with PD is challenging.

Automated mechanical peripheral stimulation (AMPS) has been recently proposed as therapy for motor and cardiovascular improvements in patients with PD. On the other hand, physical exercise has been recommended for patients with PD showing to be effective in improving physical conditioning and cognitive function.

However, the combined effects of AMPS and exercise on cardiovascular variables and functional capacity of patients with PD are still unknown.

Therefore, volunteers will be randomly allocated into two groups: 1) exercise group: will be submitted to a program of 24 exercise sessions, along with 2 weekly sessions of SHAM AMPS for 12 weeks. 2) AMPS groups: will be submitted to the program of 24 exercise sessions, along with 2 weekly sessions of AMPS during the same period.

AMPS sessions will be held prior to exercise sessions. Before and after the 12-week program, all volunteers will be submitted to assessments of cardiac autonomic control, timed up and go, and cardiopulmonary exercise testing to assess aerobic functional capacity.

The hypothesis is that the exercise program combined with AMPS therapy will provide greater improvement on the cardiovascular function and aerobic functional capacity in patients with PD, than the exercise program alone.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease
* Scoring 1 to 3 on the Hoehn and Yhar scale
* Pharmacological treatment unchanged for at least 30 days prior the study

Exclusion Criteria:

* Signs of cognitive decline, based on the results of the Mini Mental State Examination
* Cardiorespiratory, neuromuscular and musculoskeletal diseases not related to PD
* Sensory peripheral neuropathy, diabetes or any other disease known to promote autonomic dysfunction
* Changes in pharmacological treatment after inclusion in the study

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-07-30 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Timed up and go | 12 weeks
  Time spent for the participant to rise from a standard chair without armrests, walk 3 meters straight at their preferred speed, turn, walk back to the chair and sit down again. Participants will perform the test twice and the lowest total duration will be considered as the outcome
Heart rate variability | 12 weeks
  Quantification of heart rate oscillation to assess the cardiac autonomic control. This is quantified by time-domain, spectral and non-linear analysis.
Peak oxygen uptake | 12 weeks
  An incremental ramp-type protocol exercise will be used to determine the participant's aerobic capacity. Oxygen uptake will be obtained on a breath-to-breath basis during the entire exercise using an expired gas measurement system.

SECONDARY OUTCOMES:
Oxygen uptake at the ventilatory anaerobic threshold | 12 weeks
  The ventilatory anaerobic threshold will be determined from the recording of oxygen uptake and carbon dioxide production measurement during an incremental ramp-type protocol exercise using an expired gas measurement system.
24-h blood pressure | 12 weeks
  Evaluation of systolic and diastolic blood pressure during 24 hours will be recorded using an ambulatory blood pressure holter.
Sleep quality | 12 weeks
  Sleep quality will be assessed using an actigraph monitor by quantifying the sleep onset, sleep latency, sleep duration, sleep efficiency and sleep disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R Zamunér, PhD, Principal Investigator — Universidad Católica del Maule
Locations (1):
- Universidad Católica del Maule, Talca, Maule Region, Chile

IPD SHARING:
Plan to Share IPD: No
Participant data will be shared upon request at the end of the study.

REFERENCES:
- [Background] [1] Souza CFM, Almeida HCP, Souza JB, Costa PH, Silveira YSS, Bezerra JCL. A doença de Parkinson e o processo de envelhecimento motor: uma revisão da literatura. Revista de Neurociências, 2011. 19(4): p. 6.
- [Background] Barbosa MT, Caramelli P, Maia DP, Cunningham MC, Guerra HL, Lima-Costa MF, Cardoso F. Parkinsonism and Parkinson's disease in the elderly: a community-based survey in Brazil (the Bambui study). Mov Disord. 2006 Jun;21(6):800-8. doi: 10.1002/mds.20806. PMID 16482566
- [Background] Chana C P, Jimenez C M, Diaz T V, Juri C. [Parkinson disease mortality rates in Chile]. Rev Med Chil. 2013 Mar;141(3):327-31. doi: 10.4067/S0034-98872013000300007. Spanish. PMID 23900323
- [Background] Rosa JdC, Cielo CA, Cechella C. Função fonatória em pacientes com doença de Parkinson: uso de instrumento de sopro. Revista CEFAC, 2009. 11: p. 305-313.
- [Background] Teive HA, Bertucci DC Filho, Munhoz RP. Unusual motor and non-motor symptoms and signs in the early stage of Parkinson's disease. Arq Neuropsiquiatr. 2016 Oct;74(10):781-784. doi: 10.1590/0004-282X20160126. PMID 27759801
- [Background] Asahina M, Vichayanrat E, Low DA, Iodice V, Mathias CJ. Autonomic dysfunction in parkinsonian disorders: assessment and pathophysiology. J Neurol Neurosurg Psychiatry. 2013 Jun;84(6):674-80. doi: 10.1136/jnnp-2012-303135. Epub 2012 Sep 1. PMID 22942216
- [Background] Jain S, Goldstein DS. Cardiovascular dysautonomia in Parkinson disease: from pathophysiology to pathogenesis. Neurobiol Dis. 2012 Jun;46(3):572-80. doi: 10.1016/j.nbd.2011.10.025. Epub 2011 Nov 4. PMID 22094370
- [Background] Szili-Torok T, Kalman J, Paprika D, Dibo G, Rozsa Z, Rudas L. Depressed baroreflex sensitivity in patients with Alzheimer's and Parkinson's disease. Neurobiol Aging. 2001 May-Jun;22(3):435-8. doi: 10.1016/s0197-4580(01)00210-x. PMID 11378250
- [Background] Ziemssen T, Reichmann H. Treatment of dysautonomia in extrapyramidal disorders. Ther Adv Neurol Disord. 2010 Jan;3(1):53-67. doi: 10.1177/1756285609348902. PMID 21180636
- [Background] Pyatigorskaya N, Mongin M, Valabregue R, Yahia-Cherif L, Ewenczyk C, Poupon C, Debellemaniere E, Vidailhet M, Arnulf I, Lehericy S. Medulla oblongata damage and cardiac autonomic dysfunction in Parkinson disease. Neurology. 2016 Dec 13;87(24):2540-2545. doi: 10.1212/WNL.0000000000003426. Epub 2016 Nov 11. PMID 27837003
- [Background] Goldstein DS. Dysautonomia in Parkinson disease. Compr Physiol. 2014 Apr;4(2):805-26. doi: 10.1002/cphy.c130026. PMID 24715569
- [Background] Hohler AD, Zuzuarregui JR, Katz DI, Depiero TJ, Hehl CL, Leonard A, Allen V, Dentino J, Gardner M, Phenix H, Saint-Hilaire M, Ellis T. Differences in motor and cognitive function in patients with Parkinson's disease with and without orthostatic hypotension. Int J Neurosci. 2012 May;122(5):233-6. doi: 10.1080/00207454.2012.642038. Epub 2011 Dec 22. PMID 22191544
- [Background] Matinolli M, Korpelainen JT, Korpelainen R, Sotaniemi KA, Myllyla VV. Orthostatic hypotension, balance and falls in Parkinson's disease. Mov Disord. 2009 Apr 15;24(5):745-51. doi: 10.1002/mds.22457. PMID 19133666
- [Background] Sibley KM, Mochizuki G, Lakhani B, McIlroy WE. Autonomic contributions in postural control: a review of the evidence. Rev Neurosci. 2014;25(5):687-97. doi: 10.1515/revneuro-2014-0011. PMID 24854534
- [Background] Barbic F, Perego F, Canesi M, Gianni M, Biagiotti S, Costantino G, Pezzoli G, Porta A, Malliani A, Furlan R. Early abnormalities of vascular and cardiac autonomic control in Parkinson's disease without orthostatic hypotension. Hypertension. 2007 Jan;49(1):120-6. doi: 10.1161/01.HYP.0000250939.71343.7c. Epub 2006 Nov 13. PMID 17101845
- [Background] Vanderlei LC, Pastre CM, Hoshi RA, Carvalho TD, Godoy MF. Basic notions of heart rate variability and its clinical applicability. Rev Bras Cir Cardiovasc. 2009 Apr-Jun;24(2):205-17. doi: 10.1590/s0102-76382009000200018. PMID 19768301
- [Background] Hillebrand S, Gast KB, de Mutsert R, Swenne CA, Jukema JW, Middeldorp S, Rosendaal FR, Dekkers OM. Heart rate variability and first cardiovascular event in populations without known cardiovascular disease: meta-analysis and dose-response meta-regression. Europace. 2013 May;15(5):742-9. doi: 10.1093/europace/eus341. Epub 2013 Jan 30. PMID 23370966
- [Background] Kallio M, Haapaniemi T, Turkka J, Suominen K, Tolonen U, Sotaniemi K, Heikkila VP, Myllyla V. Heart rate variability in patients with untreated Parkinson's disease. Eur J Neurol. 2000 Nov;7(6):667-72. doi: 10.1046/j.1468-1331.2000.00127.x. PMID 11136353
- [Background] Allen NE, Sherrington C, Paul SS, Canning CG. Balance and falls in Parkinson's disease: a meta-analysis of the effect of exercise and motor training. Mov Disord. 2011 Aug 1;26(9):1605-15. doi: 10.1002/mds.23790. Epub 2011 Jun 14. PMID 21674624
- [Background] Peek AL, Stevens ML. Resistance training for people with Parkinson's disease (PEDro synthesis). Br J Sports Med. 2016 Sep;50(18):1158. doi: 10.1136/bjsports-2016-096311. Epub 2016 May 13. No abstract available. PMID 27467253
- [Background] Schenkman M, Hall DA, Baron AE, Schwartz RS, Mettler P, Kohrt WM. Exercise for people in early- or mid-stage Parkinson disease: a 16-month randomized controlled trial. Phys Ther. 2012 Nov;92(11):1395-410. doi: 10.2522/ptj.20110472. Epub 2012 Jul 19. PMID 22822237
- [Background] Ganesan M, Pal PK, Gupta A, Sathyaprabha TN. Treadmill gait training improves baroreflex sensitivity in Parkinson's disease. Clin Auton Res. 2014 Jun;24(3):111-8. doi: 10.1007/s10286-014-0236-z. PMID 24659140
- [Background] Barbic F, Galli M, Dalla Vecchia L, Canesi M, Cimolin V, Porta A, Bari V, Cerri G, Dipaola F, Bassani T, Cozzolino D, Pezzoli G, Furlan R. Effects of mechanical stimulation of the feet on gait and cardiovascular autonomic control in Parkinson's disease. J Appl Physiol (1985). 2014 Mar 1;116(5):495-503. doi: 10.1152/japplphysiol.01160.2013. Epub 2014 Jan 16. PMID 24436294
- [Background] Stocchi F, Sale P, Kleiner AF, Casali M, Cimolin V, de Pandis F, Albertini G, Galli M. Long-term effects of automated mechanical peripheral stimulation on gait patterns of patients with Parkinson's disease. Int J Rehabil Res. 2015 Sep;38(3):238-45. doi: 10.1097/MRR.0000000000000120. PMID 26164797
- [Background] Stuebner E, Vichayanrat E, Low DA, Mathias CJ, Isenmann S, Haensch CA. Twenty-four hour non-invasive ambulatory blood pressure and heart rate monitoring in Parkinson's disease. Front Neurol. 2013 May 15;4:49. doi: 10.3389/fneur.2013.00049. eCollection 2013. PMID 23720648
- [Background] Stuebner E, Vichayanrat E, Low DA, Mathias CJ, Isenmann S, Haensch CA. Non-dipping nocturnal blood pressure and psychosis parameters in Parkinson disease. Clin Auton Res. 2015 Apr;25(2):109-16. doi: 10.1007/s10286-015-0270-5. Epub 2015 Feb 18. PMID 25690741
- [Background] Kleiner A, Galli M, Gaglione M, Hildebrand D, Sale P, Albertini G, Stocchi F, De Pandis MF. The Parkinsonian Gait Spatiotemporal Parameters Quantified by a Single Inertial Sensor before and after Automated Mechanical Peripheral Stimulation Treatment. Parkinsons Dis. 2015;2015:390512. doi: 10.1155/2015/390512. Epub 2015 Oct 1. PMID 26495152
- [Background] Hoehn MM, Yahr MD. Parkinsonism: onset, progression and mortality. Neurology. 1967 May;17(5):427-42. doi: 10.1212/wnl.17.5.427. No abstract available. PMID 6067254
- [Background] Gelb DJ, Oliver E, Gilman S. Diagnostic criteria for Parkinson disease. Arch Neurol. 1999 Jan;56(1):33-9. doi: 10.1001/archneur.56.1.33. PMID 9923759
- [Background] Palmerini L, Mellone S, Avanzolini G, Valzania F, Chiari L. Quantification of motor impairment in Parkinson's disease using an instrumented timed up and go test. IEEE Trans Neural Syst Rehabil Eng. 2013 Jul;21(4):664-73. doi: 10.1109/TNSRE.2012.2236577. Epub 2013 Jan 1. PMID 23292821
- [Background] Shulman LM, Katzel LI, Ivey FM, Sorkin JD, Favors K, Anderson KE, Smith BA, Reich SG, Weiner WJ, Macko RF. Randomized clinical trial of 3 types of physical exercise for patients with Parkinson disease. JAMA Neurol. 2013 Feb;70(2):183-90. doi: 10.1001/jamaneurol.2013.646. PMID 23128427
- [Derived] Zelada-Astudillo N, Moreno VC, Herrera-Santelices A, Barbieri FA, Zamuner AR. Effect of the combination of automated peripheral mechanical stimulation and physical exercise on aerobic functional capacity and cardiac autonomic control in patients with Parkinson's disease: a randomized clinical trial protocol. Trials. 2021 Apr 6;22(1):250. doi: 10.1186/s13063-021-05177-w. PMID 33823928